CLINICAL TRIAL: NCT02809495
Title: Digital Application Usage for Adherence of Patients Undergoing Robotic Assisted Radical Prostatectomy Following Oncological and Postoperative Functional Outcomes
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 1-2016
Record Dates: First submitted 2016-06-17; First posted 2016-06-22 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: the Focus of This Study is to Develop an Application for Postoperative Follow-up of Patients With Prostate Cancer

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients who will use the clinical application
  Interventions: Other: use of app in smartphone
- Patients who do not make use of clinical application

INTERVENTIONS:
Other: use of app in smartphone
  Groups: Patients who will use the clinical application

SUMMARY:
Prostate cancer (PC) is the most common non-skin tumor in men and the second leading cause of death from cancer in Brazil. It accounts for 13.8% of deaths from cancer in males, similar to what happens with breast cancer in females, corresponding to 15.8% of cancer deaths in women. Mobile applications, software developed for smartphones and tablets used for many different purposes (games, communication, entertainment etc) have become important tools of mHealth (Mobile Health in Portuguese - mobile health) as they allow remote support to patients or self-promotion of health care. It has been used globally to assist in the treatment and control of various diseases such as diabetes, physical inactivity, and many others. In oncology there are several applications developed to assist in the monitoring and treatment of various cancers such as gastric and breast cancer. So far it has not developed an application for follow-up of patients with PC, to capture data on satisfaction of post-treatment patient regarding the comorbidity of surgery, and also loyalty and adherence of patients to follow-up in offices allowing a possible intervention it is done at the right time. Nor was made compared to assess whether there is benefit in using this application. Thus, the objective of this work is to develop an application for smartphones facing the postoperative follow-up of patients undergoing robotic radical prostatectomy and compare adherence to treatment compared to accompanied by traditional way patient. In addition, we will evaluate the progress of the IPSS, ICIQ and IIEF-5 compared to preoperatively in patients undergoing prostatectomy robotic radical.

ELIGIBILITY:
Inclusion Criteria:

* patients having a diagnosis of prostate cancer who are undergoing robotic radical prostatectomy for treatment of the disease and who accept to participate in the study by signing the informed consent term.

Exclusion Criteria:

* Patients who refused to participate in the study

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is a prospective randomized controlled trial. We will select prospectively 100 patients diagnosed with prostate cancer. These patients will be divided into two groups using randomisation tables (www.random.org), which are: 1. Patients who will use the clinical application (n = 50) 2. Patients who do not use the application (n = 50 - group control).
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Evaluate if the adherence of patients who use the application is greater after treatment | 24 months

IPD SHARING:
Plan to Share IPD: Undecided